CLINICAL TRIAL: NCT01378364
Title: Safety, Tolerability and Pharmacokinetics Study of Single Rising Doses of AbGn-168H Administered by Intravenous Infusion (125 μg/kg, 500 μg/kg, 1 mg/kg, 2 mg/kg) or Subcutaneous Injection (125 μg/kg, 1 mg/kg) to Healthy Male Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Groups)
Brief Title: Phase I Study of AbGn-168H in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1304.1; 2011-000713-39 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (6):
- AbGn-168H very low dose i.v. (Experimental): subject to receive a single very low dose of AbGn-168H intravenously (i.v.) or placebo
  Interventions: Drug: AbGn-168H; Drug: Placebo
- AbGn-168H low dose i.v. (Experimental): subject to receive a single low dose of AbGn-168H intravenously (i.v.) or placebo
  Interventions: Drug: AbGn-168H; Drug: Placebo
- AbGn-168H medium dose i.v. (Experimental): subject to receive a single medium dose of AbGn-168H intravenously (i.v.) or placebo
  Interventions: Drug: Placebo; Drug: AbGn-168H
- AbGn-168H high dose i.v. (Experimental): subject to receive a single high dose of AbGn-168H intravenously (i.v.) or placebo
  Interventions: Drug: Placebo; Drug: AbGn-168H
- AbGn-168H very low dose s.c. (Experimental): subject to receive a single very low dose of AbGn-168H subcutaneously (s.c.) or placebo
  Interventions: Drug: AbGn-168H; Drug: Placebo
- AbGn-168H medium dose s.c. (Experimental): subject to receive a single medium dose dose of AbGn-168H subcutaneously (s.c.) or placebo
  Interventions: Drug: Placebo; Drug: AbGn-168H

INTERVENTIONS:
Drug: AbGn-168H — single very low dose of AbGn-168H i.v.
  Arms: AbGn-168H very low dose i.v.
Drug: AbGn-168H — single low dose of AbGn-168H i.v.
  Arms: AbGn-168H low dose i.v.
Drug: Placebo — single dose of Placebo i.v.
  Arms: AbGn-168H very low dose i.v.
Drug: Placebo — single dose of Placebo i.v.
  Arms: AbGn-168H low dose i.v.
Drug: Placebo — single dose of Placebo i.v.
  Arms: AbGn-168H medium dose i.v.
Drug: Placebo — single dose of Placebo i.v.
  Arms: AbGn-168H high dose i.v.
Drug: AbGn-168H — single medium dose of AbGn-168H i.v.
  Arms: AbGn-168H medium dose i.v.
Drug: AbGn-168H — single high dose of AbGn-168H i.v.
  Arms: AbGn-168H high dose i.v.
Drug: AbGn-168H — single low dose of AbGn-168H s.c.
  Arms: AbGn-168H very low dose s.c.
Drug: Placebo — single dose of Placebo s.c.
  Arms: AbGn-168H very low dose s.c.
Drug: Placebo — single dose of Placebo s.c.
  Arms: AbGn-168H medium dose s.c.
Drug: AbGn-168H — single medium dose of AbGn-168H s.c.
  Arms: AbGn-168H medium dose s.c.

SUMMARY:
The aim of the study is to investigate safety, tolerability and pharmacokinetics of single rising doses of AbGn-168H administered by intravenous infusion or subcutaneous injection to healthy male volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)) within normal range, 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Body Mass Index (BMI) between 18.5 and 29.9 kg/m2
3. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease in the opinion of the investigator
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological and hormonal disorders
4. Chronic or relevant acute infections including hepatitis and tuberculosis, or a positive PPD skin test (5 mm or greater) at screening or within the previous 3 months
5. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
6. Use of biologic agents within 12 weeks prior to treatment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed in a descriptive way based on: Physical examination, vital sign, 12-lead ECG, clinical laboratory tests, adverse events, assessment of tolerability by investigator | 6 weeks

SECONDARY OUTCOMES:
MRT sc (mean residence time of the analyte in the body after subcutaneous injection) | 6 weeks
CL (total/apparent clearance of the analyte in plasma after intravascular administration) | 6 weeks
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | 6 weeks
V z (apparent volume of distribution during the terminal phase delta z following an intravascular dose) | 6 weeks
V z/F (apparent volume of distribution during the terminal phase delta z after extravascular administration) | 6 weeks
V ss (apparent volume of distribution at steady state following intravascular administration) | 6 weeks
C max (maximum measured concentration of the analyte in plasma) | 6 weeks
t max (time from dosing to maximum measured concentration) | 6 weeks
AUC 0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | 6 weeks
AUC 0-tz: The area under the plasma concentration-time curve over the time interval from 0 to the last timepoint at which concentrations of AbGn-168H can be measured | 6 weeks
%AUC tz-infinity: The percentage of the AUC0-infinity obtained by extrapolation from the last evaluable timepoint | 6 weeks
delta z (terminal rate constant in plasma) | 6 weeks
t 1/2 (terminal half-life of the analyte in plasma) | 6 weeks
MRT iv (mean residence time of the analyte in the body after intravenous injection or infusion) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1304.1.4901 Boehringer Ingelheim Investigational Site, Berlin, Germany